CLINICAL TRIAL: NCT00542828
Title: A Phase II Study of the Efficacy of Rabbit Anti-thymocyte Globulin (rATG) in Patients With Low and Intermediate-1 Risk Myelodysplastic Syndrome
Brief Title: Rabbit Anti-thymocyte Globulin in the Treatment of Patients With Low to Intermediate-1 Risk Myelodysplastic Syndrome
Acronym: RISE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated due to slow enrollment.
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ThymoHEM01206; 2007-002532-28 (EudraCT Number)
Record Dates: First submitted 2007-10-10; First posted 2007-10-12 (Estimated); Results first posted 2010-04-27 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-03

CONDITIONS: Myelodysplastic Syndrome (MDS)
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — thymoglobulin; Antilymphocyte Serum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Thymoglobulin (Experimental)
  Interventions: Biological: Thymoglobulin®, Rabbit Anti-thymocyte Globulin (rATG)

INTERVENTIONS:
Biological: Thymoglobulin®, Rabbit Anti-thymocyte Globulin (rATG) — All patients were to be treated with rATG 3.75 mg/kg/day administered by intravenous (IV) infusion over ≥6 hours for 5 consecutive days (cumulative dose: 18.75 mg/kg)
  Other Names: Rabbbit Anti-human thymocyte immunoglobulin

SUMMARY:
This is a Phase II, single-arm, open-label, multinational, multicenter study of rATG in patients with low or intermediate-1 risk MDS who have either failed 1 prior treatment with growth factor(s), hypomethylating agents (5-azacitidine or decitabine), or the antiangiogenic agents lenalidomide or thalidomide, or who have never been treated for MDS (i.e., treatment-naïve patients).

ELIGIBILITY:
Inclusion Criteria:

* Patient provided signed written informed consent.
* Patient had pathologically confirmed low or intermediate-1 risk MDS at the time of MDS diagnosis and at the time of screening.
* Patient had received no more than 1 prior treatment for MDS.
* Patient exhibited at least 1 hematologic cytopenia (anemia, neutropenia, or thrombocytopenia) over a period of ≥1 week.
* Patient had documentation of any prior transfusion requirements.
* Patient had an Eastern Cooperative Oncology Group (ECOG) performance score of 0, 1, or 2.
* Patient was ≥18 and ≤70 years of age at time of signing the informed consent document (ICD).
* Patient was able to adhere to study visit schedule and all other protocol requirements.
* Patient was willing to practice a medically approved method of birth control during participation in the study (at least 12 months after the last infusion of rATG) (fertile male and female patients).

Exclusion Criteria:

* Patient was pregnant or lactating.
* Patient has had prior treatment with any ATG.
* Patient has received any immunomodulatory or immunosuppressing agents (excluding steroids) <12 weeks prior to the first infusion of rATG.
* Patient has had a prior hematopoietic stem cell transplantation and/or other organ transplant.
* Patient has had a prior allergic reaction to rabbit proteins or excipients.
* Patient had any of the following subtypes of MDS: refractory anemia with ringed sideroblasts (RARS); chronic myelomonocytic leukemia (CMML) if white blood counts >13x10^9/L; or other MDS/myeloproliferative diseases (MPD).
* Patient had MDS associated with a 5q chromosomal deletion unless the patient received prior lenalidomide treatment <4 weeks prior to the first infusion of rATG.
* Patient had MDS presumed secondary to exposure to chemicals or treatment with radiotherapy or chemotherapy.
* Patient received any investigational agents within 4 weeks prior to the first infusion of rATG.
* Patient has any of the following abnormalities: serum creatinine >1.5 x upper limit of normal (ULN); aspartate transaminase (AST) and alanine transaminase (ALT) >2.5 x ULN; or serum total bilirubin >1.5 x ULN, except for unconjugated hyperbilirubinemia related to the patient's MDS.
* Patient received any treatment with non-steroidal anti-inflammatory drugs (NSAIDs) within 14 days prior to the start of treatment.
* Patient was known to be human immunodeficiency virus (HIV) positive.
* Patient had any prior diagnosis of malignancy other than MDS, unless the patient had been disease-free for at least 5 years following the completion of curative intent therapy.
* Patient had any serious medical condition (other than MDS) that would limit survival to <2 years.
* Patient had active acute or chronic infection, including cytomegaloviremia (CMV) infection or deep tissue infection.
* Patient had any other serious medical condition, uncontrolled illness (including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia), social condition, or psychiatric illness that would prevent the patient from signing the informed consent document (ICD), or would place the patient at unacceptable risk if he/she participated in the study, or that would limit compliance with study requirements.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2007-10; Primary Completion 2009-05 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (7):
- Hopital Avicenne/University, Paris, France
- Germany (2):
  - St. Johannes-Hospital Duisburg, Duisburg
  - Medizinische Hochschule Hannover, Hanover
- UMC St Radboud Centraal, Nijmegen, Netherlands
- United Kingdom (3):
  - Royal Bournemouth Hospital, Bournemouth, England
  - St. James Hospital, Leeds, England
  - King's College Hospital, London, England

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment period: 05 November 2007 through 06 May 2009. Study participants were enrolled at 7 study centers in Europe.
Pre-assignment Details: Because the study was terminated early due to slow enrollment, only 16 participants were enrolled in the study. Of these, 14 participants went on to receive treatment with Thymoglobulin.
Groups:
- Thymoglobulin: Thymoglobulin 3.75 mg/kg/day for 5 consecutive days
Period: Overall Study
Arm/Group | Thymoglobulin
Started | 16 (Number of participants enrolled in the study; of the 16 enrolled, 14 received study treatment.)
Completed | 3 (Number of participants who completed the 12-month study period.)
Not Completed | 13
Not completed — Physician Decision | 1
Not completed — Need for Prohibited Treatment | 3
Not completed — Study Prematurely Discontinued | 7
Not completed — Did Not Receive Thymoglobulin Treatment | 2

BASELINE CHARACTERISTICS:
Arm/Group | Thymoglobulin
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.4 (7.67)
Age, Customized [Number; unit: participants]
  <60 years | 10
  >=60 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 7
Race/Ethnicity, Customized [Number; unit: participants]
  Black | 1
  White | 11
  Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Achieved Hematologic Improvement (HI)
Description: This is a measure of HI in the erythroid, platelet, and neutrophil lineages. Note that HI was observed in the erythroid lineage only, which is defined as a participant who had a >=1.5 g/dL increase in hemoglobin from baseline (pretreatment value must have been <11 g/dL) and who had a relevant reduction of units of red blood cell (RBC) transfusions by an absolute number of >=4 RBC transfusions over 8 weeks as compared with the pretreatment transfusion number in the previous 8 weeks. These criteria were taken from the 2006 International Working Group criteria.
Time Frame: 12 months
Population: Number of participants analyzed includes those who received treatment with Thymoglobulin and completed follow-up efficacy assessments. However, no formal efficacy analysis was conducted due to the small sample size and early study termination.
Measure: Number; unit: participants
Arm/Group | Thymoglobulin
Number analyzed (Participants) | 13
participants | 3

2. Secondary Outcome: Number of Participants With Duration of HI
Description: This is a measure of the duration of HI for those participants who achieved HI. Duration of HI is defined as the time from confirmation of HI response to the date of first documentation of HI relapse or death due to any cause, whichever occurs first.
Time Frame: 36 months
Population: This secondary outcome measure was not formally analyzed or assessed due to the small sample size and early study termination (i.e., no study participants reached the 36-month time point).
Arm/Group | Thymoglobulin
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Participants Who Achieved Disease Remission
Description: Disease remission is defined as a participant whose best response to therapy was a complete remission or partial remission. A complete remission is defined as: bone marrow <=5% myeloblasts with normal maturation of all cell lines; persistent dysplasia noted; and peripheral blood hemoglobin >=11 g/dL, platelets >=100 x 10^9/L, neutrophils >=1.0 x 10^9/L, and blasts 0%. Partial remission is defined as: all complete remission criteria if abnormal before treatment, except bone marrow blasts decreased by >=50% over pretreatment, but still >5%; and cellularity and morphology not relevant.
Time Frame: 36 months
Population: as for outcome 2
Arm/Group | Thymoglobulin
Number analyzed (Participants) | 0

4. Secondary Outcome: Duration of Disease Remission
Description: This is a measure of the duration of overall disease remission only for those participants who achieved an overall remission. Duration of overall remission is defined as the time from first documentation of overall remission to the date of first documentation of disease relapse or death due to any cause, whichever occurs first.
Time Frame: 36 months
Population: as for outcome 2
Arm/Group | Thymoglobulin
Number analyzed (Participants) | 0

5. Secondary Outcome: Number of Participants Who Achieved Transfusion Independence
Description: This is a measure of transfusion independence, which is defined as a participant with no transfusions for a period of 8 consecutive calendar weeks after first dose. Transfusion independence was to be calculated only for those participants who had documented transfusions during the 8 weeks prior to enrollment.
Time Frame: 36 months
Population: as for outcome 2
Arm/Group | Thymoglobulin
Number analyzed (Participants) | 0

6. Secondary Outcome: Number of Participants With Duration of Transfusion Independence
Description: This is a measure of the duration of transfusion independence only for those participants who achieved transfusion independence. Duration of transfusion independence is defined as the longest period of time during which a participant requires no transfusions.
Time Frame: 36 months
Population: as for outcome 2
Arm/Group | Thymoglobulin
Number analyzed (Participants) | 0

7. Secondary Outcome: Number of Participants With a Relapse Following HI
Description: This is a measure of relapse following HI, which is defined as a participant who experiences at least one of the following: >=50% decrease from maximum response levels in granulocytes or platelets; >=1.5 g/dL reduction in hemoglobin; or transfusion dependence.
Time Frame: 36 months
Population: as for outcome 2
Arm/Group | Thymoglobulin
Number analyzed (Participants) | 0

8. Secondary Outcome: Number of Participants With a Relapse Following Overall Remission
Description: This is a measure of relapse following an overall remission only for participants who experienced either a complete or partial remission. Relapse following an overall remission is defined as a participant who meets any of the following criteria: a return to pretreatment bone marrow blast percentage; decrease of >=50% from maximum remission levels in neutrophils or platelets; reduction in hemoglobin concentration by >=1.5 g/dL from maximum remission levels; or transfusion dependence.
Time Frame: 36 months
Population: Secondary outcome measure was not formally analyzed or assessed due to early study termination and small sample size (i.e., no study participants reached the 36-month time point)
Arm/Group | Thymoglobulin
Number analyzed (Participants) | 0

9. Secondary Outcome: Number of Participants With Progression-free Survival
Description: This is a measure of a progression-free survival which is defined as the time from the participant's first dose to the date of disease progression, lost to follow-up or death due to any cause, whichever occurs first.
Time Frame: 36 months
Population: as for outcome 2
Arm/Group | Thymoglobulin
Number analyzed (Participants) | 0

10. Secondary Outcome: Number of Participants With Transformation to Acute Myeloid Leukemia
Description: This is a measure of transformation to acute myeloid leukemia only for participants who have bone marrow assessments. Transformation to acute myeloid leukemia is defined as the earliest date a participant experiences bone marrow blasts of >=20% after the start of treatment.
Time Frame: 36 months
Population: as for outcome 2
Arm/Group | Thymoglobulin
Number analyzed (Participants) | 0

11. Secondary Outcome: Number of Participants With a Cytogenetic Response
Description: This is a measure of cytogenic response for participants whose best response to therapy is a either a complete or partial cytogenetic response. A complete cytogenetic response is defined as the disappearance of the chromosomal abnormality without appearance of new ones. A partial cytogenetic response is defined as at least 50% reduction of the chromosomal abnormality.
Time Frame: 36 months
Population: as for outcome 2
Arm/Group | Thymoglobulin
Number analyzed (Participants) | 0

12. Secondary Outcome: Number of Participants With a Marrow Remission
Description: This is a measure of bone marrow complete remission for participants who experience a remission. Bone marrow complete remission is defined as a bone marrow assessment of <=5% myeloblasts and decrease by >=50% over pretreatment.
Time Frame: 36 months
Population: as for outcome 2
Arm/Group | Thymoglobulin
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected for approximately 19 months (includes all events which presented after the start of treatment through the end of study).
Description: In the event a single participant has experienced both a serious and a non-serious form of the same adverse event term, the individual has been included in the numerator ("number of affected participants") of both adverse event tables.
Arm/Group | Thymoglobulin
Serious Adverse Events (participants affected / at risk) | 7/14
Other Adverse Events (participants affected / at risk) | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Thymoglobulin (N=14)
Bradycardia (Cardiac disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Intestinal perforation (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 2
Oedema peripheral (General disorders) | 1
Pyrexia (General disorders) | 1
Serum sickness (Immune system disorders) | 2
Cellulitis (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Myositis (Musculoskeletal and connective tissue disorders) | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal failure acute (Renal and urinary disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Thymoglobulin (N=14)
Anaemia (Blood and lymphatic system disorders) | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 2
Pancytopenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Arrhythmia (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Deafness (Ear and labyrinth disorders) | 1
Conjunctival haemorrhage (Eye disorders) | 1
Eye pain (Eye disorders) | 1
Scleral hyperaemia (Eye disorders) | 1
Visual impairment (Eye disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Abdominal tenderness (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 10
Dry mouth (Gastrointestinal disorders) | 3
Dysphagia (Gastrointestinal disorders) | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1
Mouth haemorrhage (Gastrointestinal disorders) | 1
Mouth ulceration (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 5
Oral pain (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 4
Catheter site pain (General disorders) | 1
Chills (General disorders) | 3
Fatigue (General disorders) | 3
Injection site reaction (General disorders) | 1
Local swelling (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Oedema (General disorders) | 1
Oedema peripheral (General disorders) | 3
Pyrexia (General disorders) | 9
Cytokine release syndrome (Immune system disorders) | 1
Serum sickness (Immune system disorders) | 3
Central line infection (Infections and infestations) | 1
Epstein-Barr virus infection (Infections and infestations) | 1
Folliculitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 2
Staphylococcal infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 1
Blood glucose increased (Investigations) | 1
Blood lactate dehydrogenase increased (Investigations) | 1
Blood phosphorus decreased (Investigations) | 1
Blood potassium decreased (Investigations) | 1
Blood sodium increased (Investigations) | 1
Blood urine present (Investigations) | 1
Hepatic enzyme increased (Investigations) | 1
Liver function test abnormal (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 2
Protein urine present (Investigations) | 1
Weight increased (Investigations) | 2
Anorexia (Metabolism and nutrition disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1
Benign intracranial hypertension (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 6
Lethargy (Nervous system disorders) | 3
Paraesthesia (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 1
Genital ulceration (Reproductive system and breast disorders) | 1
Menorrhagia (Reproductive system and breast disorders) | 1
Menstrual disorder (Reproductive system and breast disorders) | 1
Sexual dysfunction (Reproductive system and breast disorders) | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 2
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2
Ecchymosis (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 2
Erythema (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 1
Petechiae (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1
Purpura (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 5
Rash erythematous (Skin and subcutaneous tissue disorders) | 2
Rash macular (Skin and subcutaneous tissue disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1
Skin chapped (Skin and subcutaneous tissue disorders) | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1
Swelling face (Skin and subcutaneous tissue disorders) | 1
Cardiovascular insufficiency (Vascular disorders) | 1
Flushing (Vascular disorders) | 2
Hypertension (Vascular disorders) | 3
Hypotension (Vascular disorders) | 4

LIMITATIONS AND CAVEATS:
The study was terminated early due to a slow enrollment rate; therefore, only safety data were collected from participants for 45 days following the last day of infusion (Day 5).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less